CLINICAL TRIAL: NCT02804685
Title: Effectiveness of an Exercise Protocol on Alteration of Knee Joint Position Sense in Futsal Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Guido Fabián Gómez Chiguano, Physiotherapist, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DAG Research Group
Record Dates: First submitted 2016-06-08; First posted 2016-06-17 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Proprioceptive Disorders; Knee Injuries; Athletic Injuries
MeSH Terms: conditions — Somatosensory Disorders; Knee Injuries; Athletic Injuries

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Control (No Intervention): It consists on only a regular training performance
- Experimental (Experimental): It consists on performing the protocol which includes 6 strength, agility and balance exercises together with the regular training. The exercise program has to be performed twice a week during 6 weeks
  Interventions: Other: exercise protocol

INTERVENTIONS:
Other: exercise protocol — The multi-intervention exercise protocol consists in a performance of agility, strength and balance exercises. It has to be fulfilled during 6 weeks (twice a week) before the regular training performance. The exercises should be done for almost 15 minutes approx. There will be 6 exercises in total: squat with toe raise, one-leg squats, single-leg balance (throwing a ball with a partner), vertical jumps, hamstring exercise, quick forwards and backwards sprints.
  Arms: Experimental

SUMMARY:
This research presents a randomized clinical trial which evaluates the effectiveness of an exercise protocol on the knee-joint repositioning in futsal players related to a post-match muscle fatigue. Our hypothesis is the improvement of sensation in a knee in joint position before and after the match when performing our exercise program.

ELIGIBILITY:
Inclusion Criteria:

Must have three years of experience in futsal Must be Licensed players

Exclusion Criteria:

lower limb injuries

Ages: 16 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2016-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Joint Position Sense | up to 6 weeks after the end of the intervention
  Joint Position Sense: Pictures of the knee joint repositioning of the participant are taken. The camera is placed perpendicularly 2 m from the knee joint and 65 cm from the ground. As references, 4 markers are placed in the lower extremity. The participant is seated with his feet dangling and his eyes closed. The dominant leg of the participant is passively carried by the examiner to 45 ° knee flexion. The participant is asked to maintain that position for 10 seconds. After that examiner returns the leg of the player to initial position in a passive way. The participant is then asked to change the position of the leg in an active way to the target position and maintain it for 4 seconds. After that he should return to the initial position. This exercise should be done 3 times. In each position a photograph is taken and then all of them are measured by Autocad which specifies the angles. The absolute angular error, the relative angular error and the variable angular error are measured.

SECONDARY OUTCOMES:
Vertical jump heigh | up to 6 weeks after the end of the intervention
  Vertical jump height: for this, computer software "HSC-Kinovea" must be used. To perform the jump, hands should be placed on hips and the maximum impulse should be taken with both legs in order to take off from the ground. Each participant performs 5 preparatory jumps and then another 5 jumps (as high as possible). These 5 last jumps are the ones that will be analyzed. The height of the best jump is obtained through the formula mentioned above.
  The flight time of these 5 jumps will be recorded with a camera that films 240 frames per second (Canon PowerShot SX700 HS). The analysis of the data is done with the software "Kinovea 0.8.15 for Windows" that measures the time difference between the first frame in which both feet are taking off the floor and the frame in which only one or both feet land. This measurement allows us to relate the height of each jump with muscle fatigue
Perceived exertion rate | up to 6 weeks after the end of the intervention
  Perceived exertion rate is obtained through the Borg Scale for Perceived Exertion (Borg's 6 to 10 Rating of Perceived Exertion Scale) with the aim of relating the subjective perception of the effort with objective measures of muscle fatigue. It is a discrete quantitative variable.
  Borg Scale for Perceived Exertion will be given to the participants at the end of each match. It consists of a list of numbers from 6 to 20 which are related to subjective expressions of effort (no effort: 6, extremely light: 7-8, very light: 9, light 11 moderate: 13, hard 15, very hard 17, extremely hard: 19, maximum effort: 20). The participant will be asked how they felt during this physical activity (in relation with the effort). The collected data will be related to the numeric value.

CONTACTS AND LOCATIONS:
Locations (1):
- Guido Gómez, Collado Villalba, Madrid, Spain